CLINICAL TRIAL: NCT04610970
Title: A Single-arm, Open-label, Multicenter, Phase II Clinical Trials of TQ-B3525 in Subjects With Relapse/Refractory Diffuse Large B-cell Lymphoma （DLBCL）
Brief Title: A Study of TQ-B3525 in Subjects With Relapse/Refractory Diffuse Large B-cell Lymphoma （DLBCL）
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ-B3525-II-05
Record Dates: First submitted 2020-10-26; First posted 2020-11-02 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — TQ-B3525

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ-B3525 tablets (Experimental): TQ-B3525 tablet administered orally.
  Interventions: Drug: TQ-B3525 tablets

INTERVENTIONS:
Drug: TQ-B3525 tablets — TQ-B3525 tablet administered 20mg orally, once daily in 28-day cycle.

SUMMARY:
This is a study to evaluate the efficacy and safety of TQ-B3525 in subjects with relapse/refactory diffuse large B-cell lymphoma who have received at least 2 lines of therapeutic schedules including rituximab. TQ-B3525 tablet administered 20mg orally, once daily in 28-day cycle.

ELIGIBILITY:
Inclusion Criteria:

* 1.Understood and signed an informed consent form; 2. 18 years and older, Eastern Cooperative Oncology Group(ECOG) performance status score of 0 to 2, Life expectancy ≥ 3 months; 3. Relapsed/refractory Diffuse Large B-cell lymphoma （DLBCL); 4. Has received at least two lines of previous treatment, the latest treatment confirmed no objective response, or disease progress after treatment, either of the treatment should conclude rituximab; 5. Has at least one measurable lesion; 6. Adequate organ system function; 7. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ；No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the first administration.

Exclusion Criteria:

* 1. DLBCL transformed from previously diagnosed indolent lymphoma; 2. Has central nervous system violation; 3. Has received other PI3K inhibitors or CAR-T treatments; 4. Has diagnosed and/or treated additional malignancy within 3 years prior to the first administration; 5. Has type I diabetes or uncontrolled type II diabetes; 6.Has history of interstitial lung disease; 7. Has a history of immunodeficiency diseases; 8. Has multiple factors affecting oral medication; 9.Has adverse events caused by previous therapy except alopecia that did not recover to ≤grade 1; 10. Has received systemic steroid treatment within 7 days before the first administration; 11. Has received other systemic anti-tumor medications within 4 weeks before the first administration, or still within the 5 half-life of the medication, which occurs first; 12. Has active infections within 4 weeks before the first administration; 13. Has received surgery, or unhealed wounds within 4 weeks before the first administration; 14. Has a history of autologous hematopoietic stem cell transplant within 3 months; 15. Has a history of allogeneic hematopoietic stem cell transplant; 16. Grade II or higher cardiovascular disease within 6 months before the first administration; 17. QTCF > 480ms, LVEF < 50%; 18. Urinary protein ≥ 2 +, and 24-hour urinary protein quantity>1g within 7 days; 19. Has active hepatitis B or C; 20. Has psychotropic substances abuse or a mental disorder; 21. Has other conditions that make it inappropriate for the patient to be enrolled based on investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) assessed by Independent Review Committee | Baseline up to 18 months
  Percentage of participants achieving complete response (CR) and partial response (PR) based on IRC

SECONDARY OUTCOMES:
Overall response rate (ORR) assessed by Investigator | Baseline up to 18 months
  Percentage of participants achieving complete response (CR) and partial response (PR) assessed by investigator.
Progression-free survival (PFS) | Baseline up to 18 months
  PFS was defined as the time from the date of study enrollment to the date of the first of the following events, objective disease progression or death due to any cause.
Disease control rate（DCR） | Baseline up to 18 months
  Percentage of subjects achieving complete response (CR) and partial response (PR) and stable disease (SD).
Overall Survival (OS) | Baseline up to 24 months
  OS defined as the time from the first dose to death from any cause. Survival time was censored at the date of last contact for patients who were still alive or lost to follow-up.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality